CLINICAL TRIAL: NCT01767142
Title: Feasibility Study of a Belt Applicator for Non-Invasive Fat Reduction in the Outer Thigh
Brief Title: Feasibility Study of a Belt Applicator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZA12-009
Record Dates: First submitted 2013-01-09; First posted 2013-01-14 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Body Fat Disorder
Keywords: Lipolysis; Cryolipolysis; Fat Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Outer Thigh CoolSculpting Treatment (Experimental): Treatment with the CoolSculpting System and a modified belt applicator will be performed on one outer thigh; the remaining thigh is considered the untreated control. Subjects will receive one cooling cycle applied to the thigh area intended for treatment with a protocol-defined cooling rate and duration of 120 minutes.
  Interventions: Device: The Zeltiq System with Modified Belt Applicator

INTERVENTIONS:
Device: The Zeltiq System with Modified Belt Applicator — Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
  Other Names: Cryolipolysis

SUMMARY:
Evaluate the safety and feasibility of non-invasive fat reduction in the outer thigh with a belt applicator. Applicator design and treatment parameters will be evaluated.

DETAILED DESCRIPTION:
The Zeltiq CoolSculpting System technology for cold-assisted lipolysis will be used with a modified belt applicator for the reduction of fat on the outer thigh. This is an open label, interventional, non-randomized feasibility study.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects > 18 years of age and < 65 years of age.
* Subject has clearly visible fat on intended treatment area (outer thighs), which in the investigator's opinion, may benefit from the treatment(s).
* Subject has not had weight change exceeding 10 pounds in the preceding month.
* Subject with body mass index (BMI) up to 30. BMI is defined as weight in pounds multiplied by 703 divided by the square of the height in inches.
* Subject agrees to maintain his/her weight (i.e., within 5 pounds) by not making any major changes in his/her diet or lifestyle during the course of the study.
* Subject has read and signed a written informed consent form.

Exclusion Criteria

* Subject has had a surgical procedure(s) in the area of intended treatment.
* Subject has had an invasive fat reduction procedure (e.g., liposuction, mesotherapy) in the area of intended treatment.
* Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 6 months.
* Subject needs to administer, or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
* Subject has a known history of cryoglobulinemia, cold urticaria, or paroxysmal cold hemoglobinuria.
* Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
* Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
* Subject is taking or has taken diet pills or supplements within the past month.
* Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
* Subject has an active implanted device such as a pacemaker, defibrillator, or drug delivery system
* Subject is pregnant or intending to become pregnant in the next 8 months.
* Subject is lactating or has been lactating in the past 6 months.
* Subject is unable or unwilling to comply with the study requirements.
* Subject is currently enrolled in a clinical study of any other unapproved investigational drug or device.
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bachelor, MD, Principal Investigator — Innovation Research Center
Locations (2):
- United States (2):
  - Marina Plastic Surgery, Marina del Rey, California
  - Innovation Research Center, Pleasanton, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Cryolipolysis Conformable-Surface Applicator for Nonsurgical Fat Reduction in Lateral Thighs — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4462597/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with clearly visible fat in the treatment area (outer thigh) were recruited from two clinical research sites.
Pre-assignment Details: Screening of all subjects was completed to ensure each subject met all inclusion criteria and none of the exclusion criteria. A brief medical history and exam was performed at the screening visit. All female subjects of child bearing potential were given a pregnancy test.
Units Other Than Participants: Thighs
Groups:
- Lateral Thigh Treatment Group: Treatment with the CoolSculpting System and a modified belt applicator will be performed. Non-invasive cooling is applied to one outer thigh with a protocol-defined cooling rate and duration of 120 minutes. Only one cooling cycle will be performed per subject.
Period: Overall Study
Arm/Group | Lateral Thigh Treatment Group
Started | 40; 40 Thighs (Each subject was treated on a single thigh. therefore the number of units is 40.)
Completed | 37; 37 Thighs
Not Completed | 3; 3 Thighs
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Each subject in the baseline analysis population had a unilateral CoolSculpting treatment on one outer thigh. The contralateral thigh was untreated.
Groups:
- Fat Reduction of the Lateral Thigh: Treatment with the CoolSculpting System and a modified belt applicator will be performed; non-invasive cooling is applied to the treatment area with a defined cooling rate and duration. Treatment will be applied to one (1) outer thigh.
  The Zeltiq System with Modified Belt Applicator: Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
Arm/Group | Fat Reduction of the Lateral Thigh
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 1
  Asian | 2
  Caucasian | 31
  Hispanic | 5
  Not specified | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 25.3 [20.7 to 30.4]

OUTCOME MEASURES:

1. Primary Outcome: Change in the Fat Layer of the Treated Area as Measured by Ultrasound The Change in Fat Layer Thickness in the Treated Outer Thigh
Description: For each subject, ultrasound measurements will be obtained from the treated area and the contralateral untreated control area. The change in fat layer thickness in the untreated control thigh between baseline and 16 weeks will be used to account for variation in subject body weight during the study. The fat layer thickness change in the treated area will be normalized by subtracting the change in the untreated control thigh to remove the influence of subject weight variations. The normalized value will be used to evaluate success. The result is considered the treatment effect, an absolute change, and is reported as a mean change for the study population in centimeters of fat layer reduction.
Time Frame: Baseline to 16 weeks post-final treatment
Population: The per-protocol population included all treated subjects who completed all follow-up visits and who maintained their body weight as directed by the study protocol. Six (6) subjects out of the 37 who completed the study, were excluded from the ultrasound measurement analysis because they had weight change greater than 5 pounds.
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Fat Reduction of the Lateral Thigh: Treatment with the CoolSculpting System and a modified belt applicator will be performed; non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
  The Zeltiq System with Modified Belt Applicator: Non-invasive cooling is applied to the treatment area with a defined cooling rate and duration.
Arm/Group | Fat Reduction of the Lateral Thigh
Number analyzed (Participants) | 31
cm | -0.25 (0.23)

2. Primary Outcome: Safety of the Zeltiq System and Procedure
Description: The number of device- and/or procedure related adverse events will be tabulated. Adverse event reports are collected throughout the study from the time of enrollment through the final 16 week follow-up visit. Investigators will determine whether an adverse event has a relationship to the study device or procedure.
Time Frame: Study enrollment through 16 weeks post-treatment
Population: The as-treated (safety) analysis population consists of all subjects treated in the study wherein a safety evaluation was completed. Three (3) subjects were lost to follow-up.
Measure: Number; unit: Device/procedure-related AE
Arm/Group | Fat Reduction of the Lateral Thigh
Number analyzed (Participants) | 37
Device/procedure-related AE | 1

3. Secondary Outcome: Percent of Correct Identification of Pre-treatment Photos
Description: Change in the treated vs. untreated areas will be assessed by observation of changes in surface contour and/or fat volume by an independent photo review of pre-treatment and post-treatment images of the treated areas. Reviewers will be practicing dermatologists or plastic surgeons. All reviewers will be blinded to post-treatment vs. baseline untreated area. The order in which images will be presented will be randomized; for each subject placement of the baseline, pre-treatment image will be randomized for each pair of subject images. Reviewers will be asked to select the baseline (pre-treatment) photos for each subject photo series and record selections on a data collection form. Criteria for evaluable photos for the purposes of the independent review: subject completed treatment regimen; subject has complete set of baseline photos; subject has a complete set of post-treatment photos; photos were taken using Zeltiq standard procedure.
Time Frame: Baseline and 16 weeks post-final treatment
Population: Excluded from analysis are 6 subjects who did not maintain weight within protocol requirements and 3 subjects lost to follow-up.
Measure: Count of Units; unit: Photos
Units Other Than Participants: Photos
Arm/Group | Fat Reduction of the Lateral Thigh
Number analyzed (Participants) | 31
Number analyzed (Photos) | 93
Photos | 78
Statistical Analysis 1: Comparison: Fat Reduction of the Lateral Thigh; Test type: Other; sucess proportion = 83.9, 95% CI 2-sided [74.8 to 90.7]

4. Secondary Outcome: Percentage of Participants With Satisfaction on Questionnaire Questions
Description: Subject satisfaction as assessed by questionnaires administered at 16 weeks post-treatment. The questionnaire was composed of 5-point Likert scale questions, as well as free text responses. Each question offered five choices, ranging from very favorable, somewhat favorable, neutral/not sure, unfavorable and very unfavorable responses.
Time Frame: 16 weeks post-treatment
Population: Of the forty enrolled subjects, three (3) were lost to follow-up and satisfaction questionnaires were not obtained.
Measure: Number; unit: Percent of subjects expressing satis fac
Arm/Group | Fat Reduction of the Lateral Thigh
Number analyzed (Participants) | 37
Percent of subjects expressing satis fac
  Procedure very to somewhat comfortable | 75.7
  Very visible to somewhat visible fat reduction | 86.5
  Positive overall effect | 70.3
  Very to somewhat satisfied with procedure | 86.5
  Somewhat to very different fit of clothing | 51.4
  Very likely to somewhat likely to have another tx | 97.3
  Very to somewhat likely to retreat the same area | 62.2
  Would recommend CoolSculpting to a friend | 89.19

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from enrollment until the 16-week follow-up visit.
Description: The following definition was described in the study protocol:
  Adverse events (AE) will be assessed continuously throughout the study. An adverse event is defined as any untoward medical occurrence in a subject, regardless of whether the event is related to the device or the treatment.
Arm/Group | Fat Reduction of the Lateral Thigh
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 7/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fat Reduction of the Lateral Thigh (N=40)
Seasonal cold symptoms (Infections and infestations) | 1 (1)
Injured hip (Musculoskeletal and connective tissue disorders) | 1 (1)
Runny and stuffy nose (General disorders) | 1 (1) — Subject reported symptoms of runny and stuffy nose 111 days after treatment. Condition resolved 4 days after report
Flu symptoms (Infections and infestations) | 1 (1)
Ear pain and sore throat (Infections and infestations) | 1 (1)
Pain/discomfort (General disorders) | 1 (1)
Numbness in treatment area (Skin and subcutaneous tissue disorders) | 1 (1) — Mild numbness in the treatment area persisted for 8 week post-treatment. Symptoms resolved on day 63 post-treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No